CLINICAL TRIAL: NCT03917212
Title: Non-invasive Measurement of Energy Metabolism in Patients With Primary and Secondary Mitochondrial Diseases
Brief Title: Energy Metabolism in Branched-chain Organic Acidemias
Status: Completed | Type: Observational
Sponsor: German Diabetes Center (Other)
Collaborators: University Children's Hospital, Düsseldorf (Unknown)
Responsible Party: Sponsor
Other Study IDs: MITO-MRS
Record Dates: First submitted 2019-04-09; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Energy Metabolism; Metabolic Syndrome; Insulin Resistance
Keywords: Organic acidemias; Mitochondria; Oxidative stress; Fatty liver; Dyslipidemia
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Fatty Liver; Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with propionic acidemia, isovaleric acidemia, methylmalonic acidemia
  Interventions: Other: No intervention
- Controls: Healthy humans
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention, observational study with metabolic characterisation

SUMMARY:
Energy metabolism and insulin sensitivity were assessed in a case-control study in patients with branched-chain organic acidemias.

DETAILED DESCRIPTION:
Children and adults with branched-chain organic acidemias and matched healthy humans underwent deep metabolic phenotyping using non-invasive magnetic resonance spectroscopy, oral glucose tolerance tests and measurements of leucocyte respirometry in order to assess changes in energy metabolism and insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* known branched-chain organic acidemia diagnosed by enzymatic or genetic test
* age>5 years

Exclusion Criteria:

* acute inflammatory conditions with fever, cold symptoms, gastro-intestinal infection within the last 24 hours
* contraindications for an oral glucose tolerance test such as fasting blood glucose >126 mg/dl, severe chronic gastrointestinal conditions, allergy against black currant
* contraindications for magnetic resonance tomography (MRT) such as claustrophobia, metallic implants which are not MRT compatible

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with known propionic acidemia, methylmalonic acidemia or isovaleric acidemia were enrolled as well as healthy humans of comparable age, sex and BMI
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Hepatic and skeletal muscle energy metabolism | At baseline
  Hepatic and skeletal muscle energy metabolism assessed by magnetic resonance spectroscopy

SECONDARY OUTCOMES:
Insulin sensitivity | At baseline
  Insulin sensitivity measured from oral glucose tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Professeor, Principal Investigator — German Diabetes Center; Regina Ensenauer, Professor, Principal Investigator — Children's Hospital Düsseldorf
Locations (2):
- Germany (2):
  - Department of General Pediatrics, Neonatology and Pediatric Cardiology of the University Children's Hospital Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Institute for Clinical Diabetology, German Diabetes Center, Düsseldorf, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No